CLINICAL TRIAL: NCT04308577
Title: Diet Induced Ketosis for Brain Injury - A Feasibility Study: A Ketogenic Diet With MCT Supplementation as a Potential Treatment for Brain Injury in Adults
Brief Title: Diet Induced Ketosis for Brain Injury - A Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jens Rikardt Andersen (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor-Investigator, Jens Rikardt Andersen, Associate Professor, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U Copenhagen
Record Dates: First submitted 2020-03-06; First posted 2020-03-16 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Brain Injuries; Traumatic Brain Injury; Subarachnoid Hemorrhage; Stroke; Anoxic Brain Injury; Neuroinfections
MeSH Terms: conditions — Brain Injuries; Brain Injuries, Traumatic; Subarachnoid Hemorrhage; Stroke; Hypoxia-Ischemia, Brain | interventions — Diet, Ketogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ketogenic diet with MCT (Experimental): Ketogenic Diet supplemented with MCT everyday for 6 weeks.
  Interventions: Other: Ketogenic diet with added MCT

INTERVENTIONS:
Other: Ketogenic diet with added MCT — The intervention is a ketogenic diet consisting of KetoCal 2,5:1 LQ MCT Multi Fibre (Nutricia), Liquigen (MCT)(Nutricia) and ketogenic meals provided by the hospital kitchen. The macronutrient composition of the ketogenic diet given approx.: Protein 11 E%, Carbohydrate 3 E%, Fat 86 E%.

SUMMARY:
Each year, approx. 100 patients with severe brain injury is admitted to the Clinic for Neurorehabilitation/TBI Unit, Rigshospitalet. Severe brain injury results in local oxygen deficiency and acid formation in the brain, which together destroys brain cells. The purpose of this study is to investigate whether it is possible to carry out a ketogenic diet therapy for patients with severe brain injury for six weeks. Ketosis has been shown to be neuroprotective during and after severe brain injury.

DETAILED DESCRIPTION:
Abstract

At the Department of Highly Specialized Neurorehabilitation/Traumatic Brain Injury, Rigshospitalet (satellite department at Hvidovre Hospital), approximately 100 patients (pt.) are admitted with severe brain damage every year. From 2015 to 2017, 305 pt. were admitted. Out of the 305 pt., 162pt. (53%) had traumatic brain injury (TBI), 48pt. (16%) had apoplexy, 35pt. (12%) had other diagnoses (infections, tumors and almost drowning, etc.), 20pt. (7%) had spontaneous subarachnoid hemorrhage (SAH) and 24pt. (8%) had brain damage as a result of cardiac arrest.

TBI is a leading cause of injury-related morbidity and mortality worldwide. According to the Global Burden of Disease Study (2016), there were 27,08 million new cases of TBI globally in 2016. In Denmark, there were 17.302 new cases of TBI in 2016. Clinical studies have repeatedly shown major changes in cerebral energy metabolism after TBI. The secondary brain injury leads to metabolic cellular dysfunction, cerebral edema, and a complex injury cascade. The injury spread includes processes such as inflammation, edema, free radical damage, oxidative damage, ischemic injury, cerebral glucose metabolism disorder, and ion-mediated cell damage. Much of the neurological dysfunction that occurs in acute TBI also occurs in apoplexy, SAH and cerebral ischemia.

A very important adaptive metabolic response after brain injury is the utilization of alternative cerebral energy substrates, including lactate, but also ketone bodies (KB) such as β-hydroxybutyrate (BHB) and acetoacetate (AcAc). In addition to having a central role in the regulation of cerebral energy metabolism after brain injury, KB has other important neuroprotective properties, including attenuation of oxidative stress, apoptotic cell death, and microglial activation. Increasing KB metabolism through fasting or diet-induced ketosis promotes brain resistance to stress and injury, and attenuates acute cerebral injury. Therefore, supplementing with KB, e.g. through the use of a ketogenic diet (KD) with added medium chain fatty acids (MCT), has emerged as a potential non-pharmacological neuroprotective therapy.

KD has been used for many years for the treatment of refractory epilepsy in children and studies done on adults show promising results, but experience from several studies shows major compliance issues. KD has been shown to reduce cerebral edema and apoptosis, as well as improve cerebral metabolism and behavioral outcomes in TBI rodent models, but clinical human trials on adults with TBI are lacking. Apoplexy animal models show positive effects on pathological and functional outcomes of KD intervention or exogenous ketone administration. The only human trial of KD and apoplexy shows that KD is safe and tolerated by patients with acute apoplexy. Our hypothesis is that diet-induced ketosis will reduce the extent of secondary brain damage. The purpose of the trial is to investigate whether an intervention with a ketogenic diet supplemented with MCT is feasible for 6 weeks on hospitalized pt. with severe brain damage. This is the pre-study for a controlled study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with severe acquired brain injury (TBI, stroke, SAH, anoxic brain injury or neuroinfection)
* Patients ≥ 18 years
* Understand and speak Scandinavian language
* Informed consent from patient or deputy consent if the patient is unable to give consent due to reduced state of consciousness
* Expectation of prolonged hospitalization

Exclusion Criteria:

* Contraindication to a ketogenic diet
* Dysregulated Diabetes Mellitus
* Medicated for elevated triglycerides

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2021-02-09 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Can the intervention be completed during 6 weeks hospitalization | 6 weeks
  Yes/No, % of patients with intended b-BHB (b-BHB ≥ 0,5 mmol/L) in % of intervention days
The occurrence of adverse reactions related to the ketogenic treatment, specified | 6 weeks
  % of days with adverse effects during intervention
Can patients accept the treatment | 6 weeks
  Yes/No, % of intervention days

SECONDARY OUTCOMES:
Change in Glasgow Coma Scale (GCS) | 6 weeks
  Score 3-15, higher score is better outcome
Change in Early Functional Abilities (EFA) | 6 weeks
  Total score 20-100, higher score is better outcome
Change in Functional Independence Measure (FIM) | 6 weeks
  Change in Total score 18-126, higher score is better outcome
Change in Functional Oral Intake Scale (FOIS) | 6 weeks
  Change in Score 1-7, higher score is better outcome
Change in Ranchos Los Amigos Scale (RLAS) | 6 weeks
  Change in Score 1-8, higher score is better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Maria Edwards, Student, Principal Investigator — University of Copenhagen; Jens R Andersen, MD,MPA, Study Director — University of Copenhagen
Locations (1):
- Clinic of Neurorehabilitation / TBI Unit, Rigshospitalet (Satellite Department on Hvidovre Hospital), Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Edwards MGP, Andersen JR, Curtis DJ, Riberholt CG, Poulsen I. Diet-induced ketosis in adult patients with subacute acquired brain injury: a feasibility study. Front Med (Lausanne). 2024 Mar 19;10:1305888. doi: 10.3389/fmed.2023.1305888. eCollection 2023. PMID 38571572